CLINICAL TRIAL: NCT03969641
Title: A Prospective, Randomized, Clinical Trial to Compare Adverse Birth Outcomes in Pregnant Women Receiving Quadrivalent Recombinant Influenza Vaccine (RIV4) Versus Quadrivalent Inactivated Influenza Vaccine (IIV4)
Brief Title: Safety of RIV4 Versus IIV4 in Pregnant Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); Boston Medical Center (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00101707
Record Dates: First submitted 2019-05-28; First posted 2019-05-31 (Actual); Results first posted 2022-12-27 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Safety; Adverse Event Following Immunisation; Birth Outcomes
Keywords: Vaccination; Safety; Birth outcomes; Flublok; Pregnant; Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; FluLaval

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- RIV4 (Experimental): The first recombinant inactivated influenza vaccine (RIV) using an insect baculovirus expression system and recombinant DNA technology
  Interventions: Biological: Quadrivalent Recombinant Influenza Vaccine
- IIV4 (Active Comparator): Standard inactivated influenza vaccine (IIV) manufactured involving the use of embryonated hen eggs.
  Interventions: Biological: Quadrivalent Inactivated Influenza Vaccine

INTERVENTIONS:
Biological: Quadrivalent Recombinant Influenza Vaccine — The first recombinant inactivated influenza vaccine (RIV) using an insect baculovirus expression system and recombinant DNA technology
  Other Names: Flublok Quadrivalent
  Arms: RIV4
Biological: Quadrivalent Inactivated Influenza Vaccine — Standard inactivated influenza vaccine (IIV) manufactured involving the use of embryonated hen eggs.
  Other Names: Flulaval
  Arms: IIV4

SUMMARY:
This is a prospective, randomized clinical trial. During the study, pregnant women will be randomized (1:1) to receive RIV4 or IIV4. Vaccines will be administered by licensed providers.

Prior influenza vaccine history will be verified by medical record review when possible.

Injection-site (local) and systemic reaction data will be assessed on vaccination day and during the 8 days following vaccination using either identical web-based or paper diaries, depending on study participant preference.

Maternal serum samples will be collected for antibody titers relevant to Influenza at time points that include: prior to vaccination and ~29 days post vaccination. When feasible, maternal blood at delivery and cord blood serum will be analyzed for the same antibody titers.

Pregnant women will be followed through delivery with comprehensive obstetric and neonatal outcomes obtained from medical record review for 90 days of life.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant, as determined by medical history
2. Age ≥ 18 years of age at enrollment
3. Intention of receiving influenza vaccine based on ACIP-CDC guidelines
4. Willing to provide written informed consent prior to initiation of any study procedures
5. Gestational age at vaccination ≤ 34 weeks 0 days based on reconciliation of last menstrual period and ultrasound dating. Estimated due date (EDD) and Gestational Age (GA-EDD) will be based on reconciliation of "sure" first day of the last menstrual period (LMP) and earliest dating ultrasound. If the LMP is uncertain, then the earliest dating ultrasound will be used to determine EDD and GA. If the ultrasound derived-EDD is in agreement with sure-LMP derived EDD, then the LMP-derived EDD is used to determine GA. If the ultrasound derived EDD is not in agreement with the LMP-derived EDD, the ultrasound-derived EDD is used to determine GA.
6. English or Spanish literate
7. Intention of being available for entire study period and complete all relevant study procedures, including follow-up phone calls and collection of delivery information.

Exclusion Criteria:

1. Influenza vaccine receipt during 2019-2020 or 2020-2021 influenza season prior to study enrollment.
2. Participation in this study in 2019-2020 influenza season
3. Any condition that may interfere with assessment of local injection site reactions, e.g. obscuring tattoos
4. Known or suspected immunosuppression as a result of an underlying illness or treatment
5. Use of anti-cancer chemotherapy or radiation therapy within the preceding 36 months
6. Use of oral or parenteral corticosteroids (≥ 20mg/day prednisone equivalent) or high-dose inhaled glucocorticoid for ≥ 14 consecutive days within the preceding 30 days
7. Has an active neoplastic disease (excluding non-melanoma skin cancer), a history of any hematologic malignancy, current bleeding disorder, or taking anticoagulants (a daily aspirin is acceptable)
8. Has a history of receiving immunoglobulin or other blood product (with exception of Rh immunoglobulin) within the 3 months prior to study vaccination.
9. History of febrile illness (> 100.4°F or 38°C) within the past 24 hours prior to study vaccination
10. Contraindication to IIV or RIV receipt including history of severe allergic reaction after a previous dose of any influenza vaccine; or to a vaccine component, including egg protein
11. History of Guillain-Barré syndrome within 6 weeks of a prior dose of any influenza vaccine
12. Receipt of any licensed vaccine within 7 days prior to study vaccination or intention of receiving any vaccines during 8-day post-vaccination period
13. Receipt of live vaccine during current pregnancy
14. Signs or symptoms of active preterm labor, defined as regular uterine contractions with cervical change (dilation/effacement)
15. Known multi-fetal gestation or fetal congenital anomaly, e.g. genetic abnormality or major congenital malformation based on antenatal ultrasound
16. Anyone who is already enrolled or plans to enroll in another randomized clinical trial with any drug, vaccine or medical device. Co-enrollment in observational or behavioral intervention studies are allowed at any time
17. Any condition which, in the opinion of the investigators, may pose a health risk to the participant or interfere with the evaluation of the study objectives.
18. Anyone who is a relative of any research study personnel or is an employee supervised by study staff

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geeta K Swamy, MD, Principal Investigator — Duke University; Karen R Broder, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (3):
- United States (3):
  - Boston Medical Center, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- IIV4: Subjects in this group received an intramuscular injection of 0.5mL standard quadrivalent Inactivated Influenza vaccine (IIV4), Flulaval.
- RIV4: Subjects in this group received an intramuscular injection of 0.5mL quadrivalent Recombinant Influenza Vaccine, Flublok (RIV4)
Period: Overall Study
Arm/Group | IIV4 | RIV4
Started | 193 | 191
Completed | 184 | 181
Not Completed | 9 | 10
Not completed — Lost to Follow-up | 5 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Found to be ineligible | 1 | 1
Not completed — Intrauterine fetal demise (IUFD) | 0 | 2
Not completed — Spontaneous abortion (SAB) | 2 | 1
Not completed — Elective termination | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who received study product.
Groups:
- Total: Total of all reporting groups
Arm/Group | RIV4 | IIV4 | Total
Number analyzed (Participants) | 190 | 192 | 382
Age, Customized [Median (Full Range); unit: years]
  Maternal Age | 31 [18.2 to 43.7] | 31 [18.4 to 43.8] | 31 [18.2 to 43.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 192 | 382
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 25 | 49
  Not Hispanic or Latino | 166 | 163 | 329
  Unknown or Not Reported | 0 | 4 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 63 | 63 | 126
  White | 98 | 114 | 212
  More than one race | 12 | 10 | 22
  Unknown or Not Reported | 9 | 3 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 190 | 192 | 382
Gestational Age at Enrollment [Count of Participants; unit: Participants]
  less than 20 weeks | 65 | 78 | 143
  20-34 weeks | 125 | 114 | 239
Receipt of prior influenza season vaccine [Count of Participants; unit: Participants] | 143 | 138 | 281

OUTCOME MEASURES:

1. Primary Outcome: Number of Pregnant Women Vaccinated With RIV4 Versus IIV4 With Adverse Birth Outcomes
Description: As measured by the number of women experiencing one of the following:
  * Adverse birth outcome is a composite of occurrence of at least one of the following: preterm birth, spontaneous abortion, fetal death, or neonatal death.
    * Preterm birth- born alive at less than 37 weeks and 0 days gestation
    * Spontaneous abortion (SAB)- pregnancy loss prior to 20 weeks 0 days
    * Fetal death- intrauterine death of fetus at or after 20 weeks 0 days
    * Neonatal death- infant death within first 28 days of life
Time Frame: Birth outcomes were monitored within postnatal day 28.
Population: mITT Population- any participant that was enrolled, randomized into the study, and received study vaccine
Measure: Count of Participants; unit: Participants
Arm/Group | RIV4 | IIV4
Number analyzed (Participants) | 190 | 192
Participants | 17 | 21
Statistical Analysis 1: Comparison: RIV4 vs IIV4; The null hypothesis assumes that RIV4 is inferior (i.e., RIV4 will have a higher proportion) to IIV4 in regards to the proportion of pregnant women with adverse birth outcomes; Test type: Non-Inferiority — This objective will be assessed using a one-sided noninferiority test with the alpha level set at 0.025 (1-sided) and a noninferiority margin of 10%; p < 0.0001, Cochran-Mantel-Haenszel; The upper bound of a Newcombe binomial confidence interval with Cochran-Mantel-Haenszel weighting of the difference was used, stratified by site; Difference in Proportions (RIV4 - IIV4) = -0.0214, 97.5% CI 1-sided [upper limit 0.0406] — The directional comparison was the upper bound of the confidence interval using a 10% noninferiority margin

2. Secondary Outcome: Number of Pregnant Women With Preterm Birth After RIV4 Versus IIV4 Vaccination
Description: Preterm birth is defined as born alive at less than 37 weeks and 0 days gestation.
Time Frame: Birth outcomes were monitored through 36 weeks 6 days gestation.
Population: mITT Population- any participant that was enrolled, randomized into the study, and received study vaccine
Measure: Count of Participants; unit: Participants
Arm/Group | RIV4 | IIV4
Number analyzed (Participants) | 190 | 192
Participants | 14 | 19
Statistical Analysis 1: Comparison: RIV4 vs IIV4; Preterm birth; Test type: Superiority — This proportion was compared between the RIV4 group and the IIV4 group using an exact Mantel-Haenszel statistic (calculated in Proc Logistic in SAS) in a stratified analysis by site to control for the randomization blocks at the two-sided alpha 0.05 level. The site adjusted odds ratio and corresponding 95% confidence interval for the proportion of preterm birth was also calculated; p = 0.4645, Mantel Haenszel; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.35 to 1.48]

3. Secondary Outcome: Number of Pregnant Women With Fetal or Neonatal Death After RIV4 Versus IIV4 Vaccination
Description: Fetal death is defined as intrauterine death of fetus at or after 20 weeks 0 days. Neonatal death is defined as infant death within first 28 days of life.
Time Frame: Birth outcomes were monitored through postnatal day 28.
Population: mITT Population- any participant that was enrolled, randomized into the study, and received study vaccine
Measure: Count of Participants; unit: Participants
Arm/Group | RIV4 | IIV4
Number analyzed (Participants) | 190 | 192
Participants | 2 | 0
Statistical Analysis 1: Comparison: RIV4 vs IIV4; Fetal or neonatal death; Test type: Superiority — These proportions were compared between the RIV4 group and the IIV4 group using an exact Mantel-Haenszel statistic (calculated in Proc Logistic in SAS) in a stratified analysis by site to control for the randomization blocks at the two-sided alpha 0.05 level. The site adjusted odds ratio and corresponding 95% confidence interval for the proportions of combined fetal death and neonatal death was also calculated; p = 0.2447, Mantel Haenszel; Odds Ratio (OR) = 0.00000031, 95% CI 2-sided [lower limit 0.00] (The upper limit of this CI is infinity, thus no numeric value can be provided.)

4. Secondary Outcome: Number of Pregnant Women With Spontaneous Abortion After RIV4 Versus IIV4 Vaccination
Description: Spontaneous abortion (SAB) is defined as pregnancy loss prior to 20 weeks 0 days.
Time Frame: Birth outcomes were monitored through 19 weeks 6 days gestation.
Population: mITT Population- any participant that was enrolled, randomized into the study, and received study vaccine. By definition, SAB can only occur in women that are at less than 20 weeks 0 days gestational age. All women that were at or over 20 weeks 0 days gestational age were removed from this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | RIV4 | IIV4
Number analyzed (Participants) | 62 | 72
Participants | 1 | 2
Statistical Analysis 1: Comparison: RIV4 vs IIV4; Spontaneous abortion; Test type: Superiority — This proportion was compared between the RIV4 group and the IIV4 group using an exact Mantel-Haenszel statistic in a stratified analysis by site to control for the randomization blocks at the two-sided alpha 0.05 level. The site adjusted odds ratio and corresponding 95% confidence interval for the proportion of spontaneous abortion after vaccination was also calculated. This was a subgroup analysis of only those participants vaccinated at less than 20 weeks gestational age; p = 0.6235, Mantel Haenszel; Odds Ratio (OR) = 0.50, 95% CI 2-sided [0.04 to 5.47]

5. Secondary Outcome: Number of Pregnant Women With Moderate/Severe Solicited Reactogenicity Events (Local and Systemic) Within 8 Days After Vaccination With RIV4 Versus IIV4
Description: Reactogenicity events include Injection Site Pain, Injection Site Redness, Injection Site Tenderness, Injection Site Swelling, Nausea, Vomiting, Diarrhea, Abdominal Pain, Headache, Chills/Shivering, Body Rash, Fever, Malaise (Fatigue), Myalgia (Body Aches), and Joint Pain.
Time Frame: Reactogenicity was measured for 8 days post-vaccination.
Population: mITT Population- any participant that was enrolled, randomized into the study, and received study vaccine
Measure: Count of Participants; unit: Participants
Arm/Group | RIV4 | IIV4
Number analyzed (Participants) | 190 | 192
Participants
  Injection Site Pain | 16 | 14
  Injection Site Redness | 2 | 1
  Injection Site Tenderness | 16 | 22
  Injection Site Swelling | 0 | 0
  Nausea | 7 | 13
  Vomiting | 5 | 8
  Diarrhea | 6 | 6
  Abdominal Pain | 4 | 5
  Headache | 11 | 20
  Chills/Shivering | 3 | 3
  Body Rash | 0 | 1
  Fever | 0 | 0
  Malaise (Fatigue) | 11 | 12
  Myalgia (Body Aches) | 7 | 8
  Joint Pain | 5 | 7
Statistical Analysis 1: Comparison: RIV4 vs IIV4; Injection Site Pain; Test type: Superiority — These proportions will be compared between the RIV4 group and the IIV4 group, within symptom, using an exact Mantel-Haenszel statistic (calculated in Proc Logistic in SAS) in a stratified analysis by site to control for the randomization blocks at the two-sided alpha 0.05 level; p = 0.7029, Mantel Haenszel; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.55 to 2.50]
Statistical Analysis 2: Comparison: RIV4 vs IIV4; Injection Site Redness; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.6217, Mantel Haenszel; Odds Ratio (OR) = 2.03, 95% CI 2-sided [0.18 to 22.52]
Statistical Analysis 3: Comparison: RIV4 vs IIV4; Injection Site Tenderness; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.3848, Mantel Haenszel; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.35 to 1.39]
Statistical Analysis 4: Comparison: RIV4 vs IIV4; Nausea; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.2504, Mantel Haenszel; Odds Ratio (OR) = 0.53, 95% CI 2-sided [0.21 to 1.35]
Statistical Analysis 5: Comparison: RIV4 vs IIV4; Vomiting; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.5751, Mantel Haenszel; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.20 to 1.93]
Statistical Analysis 6: Comparison: RIV4 vs IIV4; Diarrhea; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 1.0000, Mantel Haenszel; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.32 to 3.19]
Statistical Analysis 7: Comparison: RIV4 vs IIV4; Abdominal Pain; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 1.0000, Mantel Haenszel; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.21 to 3.04]
Statistical Analysis 8: Comparison: RIV4 vs IIV4; Headache; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.1326, Mantel Haenszel; Odds Ratio (OR) = 0.53, 95% CI 2-sided [0.25 to 1.13]
Statistical Analysis 9: Comparison: RIV4 vs IIV4; Chills/Shivering; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 1.0000, Mantel Haenszel; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.20 to 5.04]
Statistical Analysis 10: Comparison: RIV4 vs IIV4; Body Rash; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 1.0000, Mantel Haenszel; Odds Ratio (OR) = 0.00, 95% CI 2-sided [lower limit 0.00] (The upper limit of this CI is infinity, thus no numeric value can be provided.)
Statistical Analysis 11: Comparison: RIV4 vs IIV4; Malaise (Fatigue); Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 1.0000, Mantel Haenszel; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.39 to 2.15]
Statistical Analysis 12: Comparison: RIV4 vs IIV4; Myalgia (Body Aches); Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 1.0000, Mantel Haenszel; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.31 to 2.48]
Statistical Analysis 13: Comparison: RIV4 vs IIV4; Joint Pain; Test type: Superiority; p = 0.7704, Mantel Haenszel; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.22 to 2.29]

ADVERSE EVENTS:
Time Frame: Adverse events were collected 8 days post vaccination. Serious adverse events were collected up to 90 days post-delivery.
Description: While there were 3 cases of spontaneous abortions, these are not counted as deaths and thus are not entered under "All-Cause Mortality." These are accounted for under "Serious Adverse Events." No pregnant women died during this study. The 2 deaths in the RIV4 group were both fetal deaths.
Arm/Group | RIV4 | IIV4
All-Cause Mortality (participants affected / at risk) | 2/190 | 0/192
Serious Adverse Events (participants affected / at risk) | 14/190 | 12/192
Other Adverse Events (participants affected / at risk) | 22/190 | 22/192
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RIV4 (N=190) | IIV4 (N=192)
Opioid Dependence Relapse (General disorders) | 1 (1) | 0 (0) — Hospitalized due to relapse of opioid dependence
Vaginal Bleeding (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Preeclampsia (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 3 (3)
Spontaneous Abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Retained Products of Conception (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Resulted in a laparoscopic appendectomy
Infection (Infections and infestations) | 1 (1) | 0 (0) — Surgical site infection after laparoscopic appendectomy
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Chorioamnionitis (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Volume Overload (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Enterocolitis with abdominal abscess (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intrauterine Fetal Demise (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Preterm Premature Rupture of Membranes (PPROM) (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Bilateral Subsegmental Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Retroperitoneal hematoma (Vascular disorders) | 0 (0) | 1 (1)
Congenital Fetal Cardiac Defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Bilateral pyelectasis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Bladder outlet obstruction (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) — Including hydronephrosis due to obstruction of bladder, Hydroureter, Chronic kidney disease
ureterocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Supernumerary Digit- Left Hand (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Trisomy 21 (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
ventricular septal defect (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
Ectopic kidney (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Absent thyroid (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Short femur (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
anomalous S1 hemivertebra (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Sagittal Synostosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RIV4 (N=190) | IIV4 (N=192)
Injection Site Pain (General disorders) | 16 (16) | 14 (14)
Injection Site Tenderness (General disorders) | 16 (16) | 22 (22)
Nausea (Gastrointestinal disorders) | 7 (7) | 13 (13)
Headache (General disorders) | 11 (11) | 20 (20)
Malaise (Fatigue) (General disorders) | 11 (11) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT03969641/Prot_002.pdf
  • Statistical Analysis Plan (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT03969641/SAP_003.pdf
  • Informed Consent Form (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/41/NCT03969641/ICF_000.pdf